CLINICAL TRIAL: NCT05279768
Title: Potential Use of Umbilical Cord Mesenchymal Stem Cells and Secretoms for Infertility Therapy in Polycystic Ovary Syndrome (PCOS) Patients With Insulin Resistance.
Brief Title: Stem Cells and Secretomes for Infertility Therapy in Polycystic Ovary Syndrome (PCOS) Patients With Insulin Resistance.
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: PT. Prodia Stem Cell Indonesia (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CT/PCOS/PSI/2022
Record Dates: First submitted 2022-02-20; First posted 2022-03-15 (Actual); Last update posted 2022-09-26 (Actual); Status verified 2022-09

CONDITIONS: Polycystic Ovary Syndrome
Keywords: Umbilical Cord Mesenchymal Stem Cell; Secretome
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Secretome

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- WJ-MSCs (Experimental): Patients will be given tablet (placebo) once for 30 days, IV 0.3 million kg/bb UC-MSCs once, and nasal drop 0.5 ml/day (growth medium) for 30 days.
  Interventions: Biological: UC-MSCs
- Secretomes (Experimental): Patients will be given tablet (placebo) once for 30 days, IV placebo (NaCl 0.9%) once, and nasal drop 0.5 ml/day (Secretomes) for 30 days.
  Interventions: Biological: Secretomes
- WJ-MSCs and Secretomes (Experimental): Patients will be given tablet (placebo) once for 30 days, IV 0.3 million kg/bb UC-MSCs once, and nasal drop 0.5 ml/day (Secretomes) for 30 days.
  Interventions: Biological: UC-MSCs and Secretomes
- Control (Placebo Comparator): Patients will be given Metformin once for 30 days, IV placebo (NaCl 0.9%) once, and nasal drop 0.5 ml/day (growth medium) for 30 days.
  Interventions: Biological: Control

INTERVENTIONS:
Biological: UC-MSCs — Treatment with tablet (placebo) once for 30 days, IV 0.3 million kg/bb UC-MSCs once, and nasal drop 0.5 ml/day (growth medium) for 30 days.
  Arms: WJ-MSCs
Biological: Secretomes — Treatment with tablet (placebo) once for 30 days, IV placebo (NaCl 0.9%) once, and nasal drop 0.5 ml/day (Secretomes) for 30 days.
  Arms: Secretomes
Biological: UC-MSCs and Secretomes — Treatment with tablet (placebo) once for 30 days, IV 0.3 million kg/bb UC-MSCs once, and nasal drop 0.5 ml/day (Secretomes) for 30 days.
  Arms: WJ-MSCs and Secretomes
Biological: Control — Treatment with Metformin once for 30 days, IV placebo (NaCl 0.9%) once, and nasal drop 0.5 ml/day (growth medium) for 30 days.
  Arms: Control

SUMMARY:
The purpose of this study is to investigating the effect of Umbilical Cord Mesenchymal Stem Cell (UC-MSCs) and secretomes to insulin resistance in Polycystic Ovary Syndrome (PCOS) patients. This study has 4 arms namely UC-MSCs treatment, secretomes treatment, UC-MSCs and secretomes treatment, and control.

DETAILED DESCRIPTION:
The investigator hypothesized that PCOS patients with insulin resistance given combination of UC-MSCs and secretomes can improve their clinical and laboratory insulin resistance, haid ovulatory cycle and fertility. All group will be observed every 1,3, and 6 months after injection.

ELIGIBILITY:
Inclusion Criteria:

* PCOS patients with insulin resistance based on Rotterdam Consensus criteria, i.e. menstrual disorders (oligomenorhea/ amennorhea)
* Patients must have hiperandrogenemia clinical and laboratory proof (Ferriman Gallwey score >8)
* Patients with Free Androgen Index (FAI) >4 and ovary polycystic from USG transvaginal
* Patients with Homeostatic (HOMA) IR score ≥ 1.7

Exclusion Criteria:

* Patients who are allergic to component of WJ-MSC or Secretome.
* Patients who are not currently on hormon treatment of other resistance treatment.
* Refusing or not participating in part / all of the research process.
* Patients with positive diagnosis of hepatitis A,B,C, and HIV

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Blood serum sample | Follicular phase on day 10-12
  Sampling of the subject's blood serum will be carried out during the follicular phase on day 10-12.
Free Androgen index (FAI) | Follicular phase on day 10-12
  Free Androgen index (FAI) is calculated by total testosterone x100/SHBG
Insulin, Glucose Plasma, and Insulin Resistance | Follicular phase on day 10-12
  insulin resistance is calculated by the method: HOMA: HOMA-IR = (insulin x glucose) / 22.5 and HOMA-ß = (20 x insulin) / glucose - 3.5.
Sex Hormone Binding Globulin (SHBG) and Anti-Mullerian Hormone (AMH) | Follicular phase on day 10-12, and 1,3,6 months after stem cells
  Parameter in testing the cytokine/adipokine/hormone profile
Leptin and Adiponectine Profile | 1,3,6 months after stem cells
  Parameter in testing the cytokine/adipokine/hormone profile
TNFα, IL-1 β, IL-6, IL-10 Profile | 1,3,6 months after stem cells
  Parameter in testing the cytokine/adipokine/hormone profile

CONTACTS AND LOCATIONS:
Overall Officials: Rima Haifa, B.Sc, Study Chair — Prodia Stem Cell Indonesia
Locations (1):
- PT Prodia StemCell Indonesia, Jakarta, Indonesia